CLINICAL TRIAL: NCT04151485
Title: The Effect of the Mind/Body Program for Fertility, Hungarian Version, on Psychological Well-Being and Assisted Reproduction Technology (ART) Outcomes: A Randomized Controlled Trial
Brief Title: The Effect of the Mind/Body Program for Fertility, Hungarian Version, on Well-Being and Assisted Reproduction Outcomes
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Semmelweis University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: 83/2019
Record Dates: First submitted 2019-10-28; First posted 2019-11-05 (Actual); Last update posted 2023-05-03 (Actual); Status verified 2023-05

CONDITIONS: Infertility, Female
Keywords: female infertility; assisted reproductive technology; in vitro fertilization; intra-cytoplasmic sperm injection; pregnancy; stress; depression; anxiety; quality of life; sleep quality; circadian rhythm; mind/body
MeSH Terms: conditions — Infertility, Female; Depression; Anxiety Disorders; Sleep Initiation and Maintenance Disorders | interventions — Fertility

STUDY DESIGN:
Intervention Model Description: Mind/Body and Fertility Support Groups will be running in a parallel manner, with continuous enrollment on the basis of pre-generated random number tables. Each group will consist of 10-16 members, and run for 10 weeks. Every 11th week two new groups (one Mind/Body and one Fertility Support) will be scheduled, and so on, until the desired number of participants will be collected.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Participants, statisticians and medical staff will be blinded for intervention allocation. Since, to control the therapist variable, the two types of interventions will be done by the same person, blinding on the Care Provider's part is not possible.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mind/Body Group (Experimental): All persons allocated to the intervention group will take part in a 10-week Mind/Body skills development fertility program parallel with fertility workup and treatment.
  Interventions: Behavioral: Mind/Body Program for Fertility (Domar et al., 2011)
- Support Group (Active Comparator): All persons allocated to the comparison intervention group will take part in a 10-week fertility support program parallel with fertility workup and treatment.
  Interventions: Behavioral: Fertility Support Program

INTERVENTIONS:
Behavioral: Mind/Body Program for Fertility (Domar et al., 2011) — see Arm Description
  Arms: Mind/Body Group
Behavioral: Fertility Support Program — see Arm Description
  Arms: Support Group

SUMMARY:
Involuntary childlessness is an emotionally stressful experience; however, psychosocial counseling is typically not available in Hungarian routine fertility care. The aim of this randomized controlled trial (RCT) is to examine the effectiveness of a Mind/Body psychological fertility intervention for women in reproductive treatment. We hypothesize that participants of the Mind/Body Program for Fertility, Hungarian version, will have more favorable psychological well-being, ART outcome results than participants of the Fertility Support Groups.

DETAILED DESCRIPTION:
Involuntary childlessness imposes significant psychological burden on those affected, particularly those involved in assisted reproductive technology (ART). The reduction of psychological distress has been shown to improve the quality of life of those affected and to possibly increase chances of pregnancy. While in more developed countries psychological support is largely available in routine fertility care, it is not yet part of the Hungarian ART protocol.

In this study, the effects of a psychosocial intervention, namely, the Hungarian version of the Mind/Body Program for Fertility (Domar et al., 2011), will be tested on the psychological well-being and ART outcomes of women in reproductive treatment, in a randomized controlled pre-post design.

For this purpose, women in ART treatment will fill in screening questionnaires (on depression, anxiety, stress, etc.), and moderate to high scorers will be randomized into an intervention (Mind/Body) group (N=70) and a comparison intervention (Fertility Support) group (N=70), lasting for 10 weeks each, before and/or during an ART cycle. Both interventions will be delivered by the same clinical psychologist, listed as central contact person below, officially trained in the Mind/Body Program for Fertility by Dr. Alice Domar at Boston IVF, Waltham, Massachusetts. A smartphone application for rating subjective stress levels twice a day, from the start of the stimulation to the day of the pregnancy test, will also be administered. Additionally, whole-night sleep EEGs will be recorded.

Medical data (such as diagnosis, hormone levels, previous treatment cycles, etc.) and sociodemographic (such as age, education, etc.) and psychological variables (such as personality traits, chronotype, intelligence, etc.) as potential moderators, as well as ART outcomes will be reported. Data of respondents willing to fill in pre- and post-questionnaires but 1) not motivated to take part in the study, or 2) motivated to take part in the study, but not able to make it, will be registered but excluded from statistical analysis comparing RCT results.

ELIGIBILITY:
Inclusion Criteria: All women awaiting or undergoing infertility treatment (insemination, in vitro fertilization or intracytoplasmic sperm injection) at the Assisted Reproduction Center of the Department of Obstetrics and Gynecology at Semmelweis University, Budapest, who:

* give informed consent to participating in the study
* have sufficient knowledge of the Hungarian language

Exclusion Criteria:

* active psychotic episode
* severe depression or other major psychiatric diagnoses
* substance abuse
* eating disorders

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 177 (Actual)
Dates: Start 2019-12-15 (Actual); Primary Completion 2023-07 (Estimated); Study Completion 2023-08 (Estimated)

PRIMARY OUTCOMES:
Mean change from baseline in results on the Fertility Quality of Life tool | through study completion, an average of 2 years
  Mean change from baseline in results on the Fertility Quality of Life (FertiQoL) Core Scale, subscales and Treatment Module
Mean change from baseline in results on the SCREENIVF tool | through study completion, an average of 2 years
  Mean change from baseline in results on the SCREENIVF tool and its subscales
Clinical pregnancy | through study completion, an average of 2 years
  Rate of clinical pregnancies at post-measurement

SECONDARY OUTCOMES:
Mean change from baseline on a Likert scale measuring strength of intention to continue treatment | through study completion, an average of 2 years
  Mean change from baseline on a 10-point Likert scale measuring strength of intention to continue treatment (if first ART cycle not successful) to post-measurement

OTHER OUTCOMES:
Mean change from baseline in results on the Beck Depression Inventory | through study completion, an average of 2 years
  Mean change from baseline in results on the 21-item Beck Depression Inventory (BDI), with special attention to category change (e.g. from moderate to mild depression level, from mild to no depression)
Mean change from baseline in results on the World Health Organisation-Five Well-Being Index | through study completion, an average of 2 years
  Mean change from baseline in results on the 5-item World Health Organisation-Five Well-Being Index (WHO-5)
Mean change from baseline in results on the Spielberger State-Trait Anxiety Inventory | through study completion, an average of 2 years
  Mean change from baseline in results on the State and Trait subscales of the Spielberger State Trait Anxiety Inventory (STAI)
Mean change from baseline in results on the Short Stress Scale | through study completion, an average of 2 years
  Mean change from baseline in results on the 26-item Short Stress Scale (SSS)
Mean change from baseline in results on the Perceived Stress Scale | through study completion, an average of 2 years
  Mean change from baseline in results on the 10-item Perceived Stress Scale (PSS-10)
Mean change from baseline in results on the Life Meaning subscale of the Brief Stress and Coping Inventory | through study completion, an average of 2 years
  Mean change from baseline in results on the 7-item Life Meaning subscale of the Brief Stress and Coping Inventory (BSCI-LM)
Mean change from baseline in results on the Awareness of Mind-Body Integration and the Trusting Body Sensations subscales of the Multidimensional Assessment of Interoceptive Awareness | through study completion, an average of 2 years
  Mean change from baseline in results on the 12-item Awareness of Mind-Body Integration and the 3-item Trusting Body Sensations subscales of the Multidimensional Assessment of Interoceptive Awareness (MAIA)
Mean change from baseline in results on the Fertility Problem Stress Scales and the Coping Strategy Scales of the Copenhagen Multi-centre Psychosocial Infertility study questionnaire | through study completion, an average of 2 years
  Mean change from baseline in results on the 14-item Fertility Problem Stress Scales and the 19-item Coping Strategy Scales of the Copenhagen Multi-centre Psychosocial Infertility (COMPI) study questionnaire
Mean change from baseline in results on the Sexual Concerns subscale of the Fertility Problem Inventory | through study completion, an average of 2 years
  Mean change from baseline in results on the 8-item Sexual Concerns subscale of the Fertility Problem Inventory
Mean change from baseline in results on the Relationship Assessment Scale | through study completion, an average of 2 years
  Mean change from baseline in results on the 7-item Relationship Assessment Scale (RAS)
Mean change from baseline in results on the Pittsburgh Sleep Quality Index | through study completion, an average of 2 years
  Mean change from baseline in results on the Pittsburgh Sleep Quality Index (PSQI)
Mean change from baseline in results on the Athens Insomnia Scale | through study completion, an average of 2 years
  Mean change from baseline in results on the 8-item Athens Insomnia Scale (AIS)
Mean results on a smartphone-based Likert-scale rating momentary stress | through study completion, an average of 2 years
  Mean results on the StressFlash smartphone-based Likert-scale rating momentary stress
Number of oocytes retrieved | through study completion, an average of 2 years
  Number of oocytes retrieved at transvaginal oocyte retrieval (TVOR)
Number of oocytes fertilized | through study completion, an average of 2 years
  Number of oocytes fertilized via IVF/ICSI
Number of embryos transferred | through study completion, an average of 2 years
  Number of embryos transferred at embryo transfer (ET)

CONTACTS AND LOCATIONS:
Overall Officials: György Purebl, PhD Ass.Prof, Principal Investigator — Institute of Behavioural Sciences, Semmelweis University, Budapest
Locations (2):
- Hungary (2):
  - Assisted Reproduction Center of the Department of Obstetrics and Gynecology at Semmelweis University, Budapest
  - Institute of Behavioral Sciences at Semmelweis University, Budapest

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Domar AD, Rooney KL, Wiegand B, Orav EJ, Alper MM, Berger BM, Nikolovski J. Impact of a group mind/body intervention on pregnancy rates in IVF patients. Fertil Steril. 2011 Jun;95(7):2269-73. doi: 10.1016/j.fertnstert.2011.03.046. Epub 2011 Apr 15. PMID 21496800
- [Derived] Szigeti F J, Kazinczi C, Szabo G, Sipos M, Ujma PP, Purebl G. The clinical effectiveness of the Mind/Body Program for Infertility on wellbeing and assisted reproduction outcomes: a randomized controlled trial in search for active ingredients. Hum Reprod. 2024 Aug 1;39(8):1735-1751. doi: 10.1093/humrep/deae119. PMID 38852061